CLINICAL TRIAL: NCT03366467
Title: Effect of Sensory Adapted Dental Environment on Children's Behavior During Dental Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The clinic no longer have sensory adapted environment equipment
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Avia Fux, pediatric dentist, Hadassah Medical Organization
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 0469-17-HMO
Record Dates: First submitted 2017-11-27; First posted 2017-12-08 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Child Behavior
Keywords: dental treatment; sensory adapted environment
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Intervention Model Description: The participants will be randomly assigned into two groups. Group 1 will initially be treated under SADE (Time 1) and receive RDE on the second encounter (Time 2). For the second group, the procedure is reversed (RDE at Time 1 and SADE at Time 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SADE first (Experimental): SADE first will initially be treated under SADE (Time 1) and receive RDE on the second encounter (Time 2)
  Interventions: Other: SADE; Other: RDE
- RDE first (Experimental): RDE first will initially be treated under RDE (Time 1) and receive SADE on the second encounter (Time 2)
  Interventions: Other: SADE; Other: RDE

INTERVENTIONS:
Other: SADE — The SADE: the sensory stimuli addressed are visual and auditory, as follows: (i) Visual sensation. All ceiling fluorescent lighting are removed. The adapted lighting consisted of slow-moving, repetitive visual color effects created by a projector, in the child's visual field. (ii) Auditory stimuli include rhythmic music, which was heard via loudspeakers.
Other: RDE — The RDE utilized fluorescent lighting on the ceiling, without special visual effects and without music stimulation.

SUMMARY:
The objective of the present study is to determine the effect of sensory adapted dental environment (SADE) in healthy children during a routine dental restorative treatment. The hypothesis is that the SADE would have a favorable effect in calming the subjects during dental treatment.

the study is a random cross-over design. The participants will be randomly assigned into two groups. Group 1 will initially be treated under SADE (Time 1) and receive regular dental environment (RDE) on the second encounter (Time 2). For the second group, the procedure is reversed (RDE at Time 1 and SADE at Time 2).

DETAILED DESCRIPTION:
* Dental treatment- will include restorations, crowns, pulp treatment, with local anesthesia. The use of oral/inhaled sedation will be decided according to the patient's behavior and cooperation assessment.
* Dental settings- The SADE: the sensory stimuli addressed are visual and auditory, as follows: (i) Visual sensation. All ceiling fluorescent lighting are removed. The adapted lighting consisted of slow-moving, repetitive visual color effects created by a projector, in the child's visual field. (ii) Auditory stimuli include rhythmic music, which was heard via loudspeakers. The RDE utilized fluorescent lighting on the ceiling, without special visual effects and without music stimulation.
* Instruments- 1) the children will be observed during the treatments. The observer will code all behaviors according to the Houpt Scale used for rating patient behavior during treatment. In addition, the examiner will count the number and duration (in minutes) of the anxious behavior (crying and movements). Because of the nature of the study (one environment with sensory adaptation and the other without), the observer cannot be blind to the treatment environment. 2) Physiologic arousal states, evaluated by the assessment of EDA (Mindlife Co, Jerusalem, Israel). Changes in the electrical conductance of the skin are a sensitive way of monitoring autonomic responses to external stimuli.

ELIGIBILITY:
Inclusion Criteria:

* ASA1
* Needs at least 2 similar dental treatment appointments

Exclusion Criteria:

* Needs only one dental treatment

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Physiologic arousal states | Data will be reported through study completion, an average of 2 years
  Evaluated by palmar electrodermal activity (EDA) during dental treatment

SECONDARY OUTCOMES:
Houpt Scale | Data will be reported through study completion, an average of 2 years
  Rating patient behavior during treatment according to Houpt scale. The Houpt scale is a tool used to assess a child's behavior during dental sedation according to specific categories and scores including: sleep (1-awake, 2-drowsy, disoriented), movement (1-violent, 2-continuous, 3-controllable, 4-no movement), cry (1-hysterical, 2-continuous, 3-intermittent, 4-no cry), and overall behavior (1-treatment aborted, 2-poor, 3-regular, 4-good, 5-very good, 6-excellent).
Anxious behavior-number | Data will be reported through study completion, an average of 2 years
  Examiner will count the number of the anxious behavior episodes (crying and movements) during dental treatment.
Anxious behavior-duration | Data will be reported through study completion, an average of 2 years
  Examiner will count the duration, in minute, of the anxious behavior (crying and movements) during dental treatment..